CLINICAL TRIAL: NCT02448719
Title: A Randomized, Single-Center, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Oral Dose of TAK-792 in Healthy Subjects
Brief Title: Single-Dose Phase 1 Study of TAK-792
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-792-1001; U1111-1170-1571 (Other: WHO); JapicCTI-152897 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Healthy Male Adults Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- Cohort 1-active (Experimental): Single oral administration of TAK-792 30 milligram (mg) in Japanese participants
  Interventions: Drug: TAK-792 30 mg
- Cohort 1-placebo (Placebo Comparator): Single oral administration of TAK-792 30 mg placebo in Japanese participants
  Interventions: Drug: TAK-792 30 mg placebo
- Cohort 2-active (Experimental): Single oral administration of TAK-792 100 mg in Japanese participants
  Interventions: Drug: TAK-792 100 mg
- Cohort 2-placebo (Placebo Comparator): Single oral administration of TAK-792 100 mg placebo in Japanese participants
  Interventions: Drug: TAK-792 100 mg placebo
- Cohort 3-active (Experimental): Single oral administration of TAK-792 250 mg in Japanese participants
  Interventions: Drug: TAK-792 250 mg
- Cohort 3-placebo (Placebo Comparator): Single oral administration of TAK-792 250 mg placebo in Japanese participants
  Interventions: Drug: TAK-792 250 mg placebo
- Cohort 4-active (Experimental): Single oral administration of TAK-792 500 mg in Japanese and Caucasian participants
  Interventions: Drug: TAK-792 500 mg
- Cohort 4-placebo (Placebo Comparator): Single oral administration of TAK-792 500 mg placebo in Japanese and Caucasian participants
  Interventions: Drug: TAK-792 500 mg placebo
- Cohort 5-active (Experimental): Single oral administration of TAK-792 750 mg in Japanese and Caucasian participants
  Interventions: Drug: TAK-792 750 mg
- Cohort 5-placebo (Placebo Comparator): Single oral administration of TAK-792 750 mg placebo in Japanese and Caucasian participants
  Interventions: Drug: TAK-792 750 mg placebo
- Cohort 6-active (Experimental): Single oral administration of TAK-792 1250 mg in Japanese and Caucasian participants
  Interventions: Drug: TAK-792 1250 mg
- Cohort 6-placebo (Placebo Comparator): Single oral administration of TAK-792 1250 mg placebo in Japanese and Caucasian participants
  Interventions: Drug: TAK-792 1250 mg placebo

INTERVENTIONS:
Drug: TAK-792 30 mg — TAK-792 30 mg was administered in the morning after a fast.
  Arms: Cohort 1-active
Drug: TAK-792 30 mg placebo — TAK-792 30 mg placebo was administered in the morning after a fast.
  Arms: Cohort 1-placebo
Drug: TAK-792 100 mg — TAK-792 100 mg was administered in the morning after a fast.
  Arms: Cohort 2-active
Drug: TAK-792 100 mg placebo — TAK-792 100 mg placebo was administered in the morning after a fast.
  Arms: Cohort 2-placebo
Drug: TAK-792 250 mg — TAK-792 250 mg was administered in the morning after a fast.
  Arms: Cohort 3-active
Drug: TAK-792 250 mg placebo — TAK-792 250 mg placebo was administered in the morning after a fast.
  Arms: Cohort 3-placebo
Drug: TAK-792 500 mg — TAK-792 500 mg was administered in the morning after a fast or after breakfast.
  Arms: Cohort 4-active
Drug: TAK-792 500 mg placebo — TAK-792 500 mg placebo was administered in the morning after a fast or after breakfast.
  Arms: Cohort 4-placebo
Drug: TAK-792 750 mg — TAK-792 750 mg was administered in the morning after a fast.
  Arms: Cohort 5-active
Drug: TAK-792 750 mg placebo — TAK-792 750 mg placebo was administered in the morning after a fast.
  Arms: Cohort 5-placebo
Drug: TAK-792 1250 mg — TAK-792 1250 mg was administered in the morning after a fast.
  Arms: Cohort 6-active
Drug: TAK-792 1250 mg placebo — TAK-792 1250 mg placebo was administered in the morning after a fast.
  Arms: Cohort 6-placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability profile of TAK-792 when administered as a single oral dose in healthy Japanese and Caucasian male participants.

DETAILED DESCRIPTION:
This study will be double-blind and placebo-controlled to avoid subjective bias in the assessment of safety and tolerability of TAK-792. Sentinel dosing will be used in the first cohort (cohort 1) to ensure adequate safety and tolerability evaluation prior to administering TAK-792 to the remainder of participants within the cohort. The dose escalation to the next cohort for Cohorts 2 to 6 will occur after full review of safety and tolerability of the current cohort, and available pharmacokinetic data up to 24 hours in the preceding cohorts. The planned dose levels are 30, 100, 250, 500, 750 and 1250 mg, to be administered in the morning after a fast of at least 10 hours.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is a healthy male of Japanese descent (born to Japanese parents and grandparents) or Caucasian descent (born to Caucasian parents and grandparents).
4. The participant is aged 20 to 45 years, inclusive, at the time of informed consent.
5. The participant weighs at least 50 kilogram (kg) and has a body mass index (BMI) between 18.5 kilogram per square meter (kg/m^2) and 25.0 kg/m^2 for Japanese, BMI between 18.5 kg/m^2 and 30.0 kg/m^2 for Caucasian, inclusive at Screening and Day -1.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.

Exclusion Criteria:.

1. The participant has received any investigational compound within 16 weeks (112 days) prior to the dose of study medication.
2. The participant is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
3. The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
4. The participant has a positive urine drug result for drugs of abuse at Screening.
5. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
6. Participant has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products table.
7. The participant intends to donate sperm during the course of this study or for 12 weeks thereafter.
8. Participant has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash.
9. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis frequent [more than once per week] occurrence of heartburn, or any surgical intervention [eg, cholecystectomy]).
10. Participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
11. Participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at Screening.
12. Participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening.
13. The participant has poor peripheral venous access.
14. The participant has undergone whole blood collection of at least 200 milliliter (mL) within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of study drug administration.
15. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of study drug administration.
16. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of study drug administration.
17. Participant has a Screening abnormal (clinically significant) electrocardiogram (ECG).
18. Participant has abnormal Screening laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than (>)1.5 the upper limits of normal.
19. Participant who, in the opinion of the investigator or sub-investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (1):
- Kagoshima, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 27 May 2015 to 28 January 2016.
Pre-assignment Details: Healthy Japanese participants received TAK-792 or placebo in Cohort 1a (30 milligram [mg]), Cohort 2a (100 mg), Cohort 3a (250 mg), Cohort 4a (500 mg), Cohort 5a (750 mg), and Cohort 6a (1250 mg). Healthy Caucasian participants received TAK-792 or placebo in Cohort 4b (500 mg), Cohort 5b (750 mg) and Cohort 6b (1250 mg).
Groups:
- Cohort 1a-6a: Placebo: TAK-792 placebo-matching tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 1a: TAK-792 30 mg: TAK-792 30 mg, tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 2a: TAK-792 100 mg: TAK-792 100 mg, tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 3a: TAK-792 250 mg: TAK-792 250 mg, tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 4a: TAK-792 500 mg: TAK-792 500 mg, tablets, orally, once in fasted state (4a-1) on Day 1 of 5-day treatment period, in Japanese participants. Participants also received same medication later in fed state (4a-2) on Day 1 of another 5-day treatment period.
- Cohort 5a: TAK-792 750 mg: TAK-792 750 mg, tablets, orally in fasted state (5a-1), once on Day 1 of 5-day treatment period, in Japanese participants. Participants also received same medication later in fasted state (5a-2) on Day 1 of another 5-day treatment period.
- Cohort 6a: TAK-792 1250 mg: TAK-792 1250 mg, tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 4b-6b: Placebo: TAK-792 placebo-matching tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Caucasian participants.
- Cohort 4b: TAK-792 500 mg: TAK-792 500 mg, tablets, orally, once in fasted state (4b-1) on Day 1 of 5-day treatment period, in Caucasian participants. Participants also received same medication later in fed state (4b-2) on Day 1 of another 5-day treatment period.
- Cohort 5b: TAK-792 750 mg: TAK-792 750 mg, tablets, orally in fasted state (5b-1), once on Day 1 of 5-day treatment period, in Caucasian participants. Participants also received same medication later in fasted state (5b-2) on Day 1 of another 5-day treatment period.
- Cohort 6b: TAK-792 1250 mg: TAK-792 1250 mg, tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Caucasian participants.
Period: Overall Study
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a: TAK-792 500 mg | Cohort 5a: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4b-6b: Placebo | Cohort 4b: TAK-792 500 mg | Cohort 5b: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic (PK) analysis set included all participants who had received the study drug and met the essential requirements defined in the study protocol without any critical protocol violations, and in whom PK assessment was possible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a: TAK-792 500 mg | Cohort 5a: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4b-6b: Placebo | Cohort 4b: TAK-792 500 mg | Cohort 5b: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 71
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 71
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 0 | 0 | 0 | 0 | 47
  Caucasian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
Region of Enrollment [Number; unit: participants]
  Japan | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 71
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 6 | 3 | 4 | 4 | 4 | 3 | 3 | 4 | 4 | 5 | 2 | 42
  Ex-Smoker | 6 | 3 | 2 | 2 | 1 | 3 | 3 | 2 | 2 | 1 | 4 | 29
Alcohol Classification [Count of Participants; unit: Participants]
  Drank a few days per week | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 5
  Drank a few days per month | 6 | 3 | 4 | 4 | 3 | 3 | 4 | 4 | 4 | 6 | 5 | 46
  Did not drink | 4 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 0 | 0 | 20
Caffeine Classification [Count of Participants; unit: Participants]
  Caffeine Consumption | 3 | 3 | 4 | 0 | 3 | 2 | 2 | 2 | 3 | 3 | 1 | 26
  No Caffeine Consumption | 9 | 3 | 2 | 6 | 2 | 4 | 4 | 4 | 3 | 3 | 5 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to Day 8
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 4a-1: TAK-792 500 mg: TAK-792 500 mg, tablets, orally in fasted state, once on Day 1 of 5 days treatment period, in Japanese participants.
- Cohort 5a-1: TAK-792 750 mg: TAK-792 750 mg, tablets, orally in fasted state, once on Day 1 of 5 days treatment period, in Japanese participants.
- Cohort 4a-2: Placebo: TAK-792 placebo-matching tablets, orally in fed state, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 4a-2: TAK-792 500 mg: TAK-792 500 mg, tablets, orally in fed state, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 5a-2: Placebo: TAK-792 placebo-matching tablets, orally in fasted state, fast state was broken immediately after the drug administration, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 5a-2: TAK-792 750 mg: TAK-792 750 mg, tablets, orally in fasted state, fast state was broken immediately after the drug administration, once on Day 1 of 5-day treatment period, in Japanese participants.
- Cohort 4b-1 - 6b: Placebo: TAK-792 placebo-matching tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Caucasian participants.
- Cohort 4b-1: TAK-792 500 mg: TAK-792 500 mg, tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Caucasian participants.
- Cohort 5b-1: TAK-792 750 mg: TAK-792 750 mg, tablets, orally in fasted state, once on Day 1 of 5-day treatment period, in Caucasian participants.
- Cohort 4b-2: Placebo: TAK-792 placebo-matching tablets, orally in fed state, once on Day 1 of 5-day treatment period, in Caucasian participants.
- Cohort 4b-2: TAK-792 500 mg: TAK-792 500 mg, tablets, orally in fed state, once on Day 1 of 5-day treatment period, in Caucasian participants.
- Cohort 5b-2: Placebo: TAK-792 placebo-matching tablets, orally in fasted state, fast state was broken immediately after the drug administration, once on Day 1 of 5-day treatment period, in Caucasian participants.
- Cohort 5b-2: TAK-792 750 mg: TAK-792 750 mg, tablets, orally in fasted state, fast state was broken immediately after the drug administration, once on Day 1 of 5-day treatment period, in Caucasian participants.
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1 - 6b: Placebo | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 2 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 2 | 6
percentage of participants | 16.7 | 16.7 | 0.0 | 33.3 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 50.0 | 33.3 | 0.0 | 33.3 | 50.0 | 16.7 | 0.0 | 16.7

2. Primary Outcome: Number of Participants With TEAE Related to Vital Signs
Description: Vital signs included body temperature (infra-axillary measurement), supine blood pressure (systolic and diastolic) after the participant has rested for at least 5 minutes, respiratory rate, and pulse (beats per minute [bpm]).
Time Frame: Baseline up to Day 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1 - 6b: Placebo | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 2 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With TEAE Related to Body Weight
Time Frame: Baseline up to Day 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1 - 6b: Placebo | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 2 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With TEAE Related to Electrocardiograms (ECG)
Time Frame: Baseline up to Day 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1 - 6b: Placebo | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 2 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs Related to Laboratory Tests
Description: Reported TEAE Related to Laboratory Tests are following; Occult blood positive, Alanine aminotransferase increased, Aspartate aminotransferase increased, Blood bilirubin increased, Blood creatine phosphokinase increased, Blood glucose increased, Blood triglycerides increased, Blood urine present, Protein urine present, and White blood cell count increased.
Time Frame: Baseline up to Day 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1 - 6b: Placebo | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 2 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 2 | 6
Participants
  Occult blood positive | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood glucose increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood triglycerides increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood urine present | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Protein urine present | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  White blood cell count increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With TEAE Related to Gastrointestinal Symptom Rating Scale (GSRS)
Description: The gastrointestinal (GI) symptoms (abdominal pain, heartburn, acid regurgitation, hunger pains, nausea, borborygmus, abdominal distension, eructation, increased flatus, constipation, diarrhoea, loose stools, hard stools, urgent need for defecation, and feeling of incomplete evacuation) using GSRS questionnaires at each assessment point. The GSRS a 15-item self-administered questionnaire that assesses the impact of GI symptoms during the past week on a scale from 1 (no discomfort at all) to 7 (very severe discomfort). Possible overall scores range from 1 to 7, with lower scores indicating a better quality of life with respect to GI symptoms. TEAEs related to GSRS were reported as follows: Diarrhoea, Constipation, Faeces hard, and Faeces soft.
Time Frame: Baseline up to Day 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1 - 6b: Placebo | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 2 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 2 | 6
Participants
  Diarrhoea | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Faeces hard | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Faeces soft | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: AUC(0-96): Area Under the Plasma Concentration-time Curve From Time 0 to 96 Hours Postdose for TAK-792F and Its Metabolites M-I and M-II
Time Frame: Day 1: pre-dose and at multiple timepoints (0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 hours post dose; up to 96 hours) post-dose
Population: PK analysis set included all participants who had received the study drug and met the essential requirements defined in the study protocol without any critical protocol violations, and in whom PK assessment was possible.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL)
  TAK-792F | 47.34 (24.7) | 350.0 (15.7) | 521.3 (24.6) | 770.6 (36.4) | 998.5 (53.2) | 1988.0 (40.8) | 357.2 (44.5) | 898.6 (28.5) | 610.5 (28.3) | 622.5 (51.8) | 557.0 (53.9) | 485.6 (31.5) | 558.2 (50.3)
  M-I | 6.765 (25.9) | 84.01 (40.8) | 63.94 (51.7) | 128.1 (27.7) | 167.6 (43.1) | 424.2 (41.9) | 79.70 (34.2) | 190.5 (51.3) | 133.6 (39.5) | 224.0 (34.7) | 407.9 (40.7) | 97.17 (36.6) | 177.6 (41.0)
  M-II | 422.5 (22.1) | 1324.0 (45.7) | 2658.0 (57.9) | 3192.0 (56.3) | 4909.0 (56.2) | 5086.0 (78.9) | 3237.0 (66.9) | 5483.0 (54.8) | 4824.0 (38.4) | 6261.0 (51.1) | 15430.0 (26.7) | 4813.0 (32.9) | 7156.0 (17.4)

8. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-792F and Its Metabolites M-I and M-II
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL
  TAK-792F | 46.45 (24.2) | 346.6 (15.4) | 517.4 (24.8) | 767.8 (36.6) | 995.9 (53.4) | 1980.0 (41.0) | 356.2 (44.6) | 891.9 (28.7) | 608.4 (28.4) | 619.2 (51.8) | 554.9 (54.1) | 481.9 (31.8) | 553.6 (50.9)
  M-I | 5.912 (31.6) | 80.78 (39.6) | 61.32 (52.1) | 119.6 (22.4) | 160.5 (42.8) | 388.6 (43.3) | 74.37 (34.7) | 182.1 (53.2) | 127.6 (41.4) | 214.3 (36.5) | 386.8 (42.4) | 92.89 (37.9) | 169.5 (41.9)
  M-II | 392.0 (24.3) | 1246.0 (46.0) | 2302.0 (57.0) | 3039.0 (52.9) | 4470.0 (59.3) | 4352.0 (71.2) | 3193.0 (68.0) | 5319.0 (56.3) | 4554.0 (41.2) | 6030.0 (54.0) | 15430.0 (26.7) | 4683.0 (34.9) | 6836.0 (17.9)

9. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-792F and Its Metabolites M-I and M-II
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  TAK-792F | 8.916 (24.2) | 59.17 (29.7) | 85.12 (21.1) | 113.2 (62.9) | 140.6 (52.6) | 267.5 (51.8) | 57.85 (48.7) | 136.4 (40.8) | 88.44 (19.8) | 97.62 (59.3) | 96.99 (47.0) | 72.22 (38.2) | 86.20 (40.9)
  M-I | 1.707 (30.8) | 13.40 (21.5) | 8.786 (29.9) | 14.0 (17.1) | 17.13 (42.6) | 37.54 (51.4) | 8.401 (34.5) | 21.92 (49.3) | 14.65 (31.7) | 21.73 (34.7) | 25.15 (28.8) | 12.86 (24.5) | 20.04 (34.3)
  M-II | 27.36 (58.9) | 87.07 (57.9) | 110.4 (70.4) | 105.2 (19.1) | 187.2 (24.0) | 213.6 (60.6) | 150.2 (27.1) | 218.9 (60.3) | 134.7 (33.4) | 193.7 (25.4) | 307.5 (10.5) | 186.4 (42.0) | 352.3 (39.8)

10. Secondary Outcome: Tmax: Time to Reach the Cmax for TAK-792F and Its Metabolites M-I and M-II
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
hours
  TAK-792F | 1.7500 (24.2) [1.500 to 4.000] | 2.5000 (29.7) [1.500 to 4.000] | 2.5000 (21.1) [1.500 to 4.000] | 2.0000 (62.9) [1.500 to 4.000] | 4.0000 (52.6) [3.000 to 4.000] | 4.0000 (51.8) [3.000 to 6.000] | 3.0000 (48.7) [1.000 to 4.000] | 3.5000 (40.8) [3.000 to 4.000] | 3.0000 (19.8) [3.000 to 6.000] | 4.0000 (59.3) [3.000 to 4.000] | 3.5000 (47.0) [2.000 to 4.000] | 3.0000 (38.2) [1.500 to 8.000] | 3.5000 (40.9) [2.000 to 4.000]
  M-I | 1.5000 (30.8) [1.000 to 3.000] | 2.0000 (21.5) [1.500 to 8.000] | 1.7500 (29.9) [1.500 to 4.000] | 6.0000 (17.1) [1.500 to 8.000] | 3.5000 (42.6) [1.500 to 8.000] | 4.0000 (51.4) [3.000 to 8.000] | 3.0000 (34.5) [1.500 to 6.000] | 3.5000 (49.3) [3.000 to 16.000] | 2.5000 (31.7) [1.000 to 6.000] | 5.0000 (34.7) [1.000 to 8.000] | 6.0000 (28.8) [2.000 to 10.000] | 4.0000 (24.5) [2.000 to 8.000] | 5.0000 (34.3) [3.000 to 10.000]
  M-II | 9.0000 (58.9) [6.000 to 12.000] | 11.0000 (57.9) [8.000 to 24.000] | 14.0000 (70.4) [10.000 to 24.000] | 16.0000 (19.1) [12.000 to 24.000] | 30.0000 (24.0) [8.000 to 48.000] | 24.0000 (60.6) [24.000 to 48.000] | 24.0000 (27.1) [10.000 to 24.000] | 16.0000 (60.3) [16.000 to 24.000] | 24.0000 (33.4) [12.000 to 24.000] | 20.0000 (25.4) [16.000 to 36.000] | 42.0000 (10.5) [24.000 to 48.000] | 16.0000 (42.0) [10.000 to 24.000] | 16.0000 (39.8) [10.000 to 24.000]

11. Secondary Outcome: Urinary Excretion Ratio of TAK-792F and Its Metabolites M-I and M-II as Percentage of TAK-792 Dose From 0 to 96 Hours Postdose
Time Frame: Day 1: pre-dose and at multiple timepoints (6, 12, 24, 36, 48, 72, 96 hours post dose; up to 96 hours) post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage (%) of dose
Arm/Group | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
percentage (%) of dose
  TAK-792F | 0.4903 (0.12275) [1.500 to 4.000] | 1.0367 (0.18525) [1.500 to 4.000] | 0.6143 (0.19055) [1.500 to 4.000] | 0.5128 (0.13384) [1.500 to 4.000] | 0.4733 (0.21291) [3.000 to 4.000] | 0.5477 (0.24886) [3.000 to 6.000] | 0.2500 (0.12329) [1.000 to 4.000] | 0.4484 (0.19575) [3.000 to 4.000] | 0.3955 (0.10436) [3.000 to 6.000] | 0.2830 (0.16074) [3.000 to 4.000] | 0.1715 (0.07766) [2.000 to 4.000] | 0.2755 (0.08876) [1.500 to 8.000] | 0.2870 (0.14673) [2.000 to 4.000]
  M-I | 1.5667 (0.35517) [1.000 to 3.000] | 1.9150 (0.72213) [1.500 to 8.000] | 1.8183 (1.03695) [1.500 to 4.000] | 1.4910 (0.62949) [1.500 to 8.000] | 0.9552 (0.56474) [1.500 to 8.000] | 1.2642 (0.51113) [3.000 to 8.000] | 0.6604 (0.24546) [1.500 to 6.000] | 1.0155 (0.62088) [3.000 to 16.000] | 1.3317 (0.85211) [1.000 to 6.000] | 1.1630 (0.25033) [1.000 to 8.000] | 1.1442 (0.31888) [2.000 to 10.000] | 0.6330 (0.32789) [2.000 to 8.000] | 0.7723 (0.24873) [3.000 to 10.000]
  M-II | 52.2833 (9.37452) [6.000 to 12.000] | 25.4567 (14.21242) [8.000 to 24.000] | 35.1333 (18.44361) [10.000 to 24.000] | 21.9300 (12.94284) [12.000 to 24.000] | 18.1750 (7.30395) [8.000 to 48.000] | 15.2100 (11.38256) [24.000 to 48.000] | 20.0120 (12.08593) [10.000 to 24.000] | 24.9333 (13.03927) [16.000 to 24.000] | 31.8350 (17.55999) [12.000 to 24.0000] | 24.4667 (13.80343) [16.000 to 36.000] | 39.4167 (9.21421) [24.000 to 48.000] | 22.5383 (15.47892) [10.000 to 24.000] | 26.7167 (8.29516) [10.000 to 24.000]

12. Secondary Outcome: AUC(0-2.5): Area Under the Plasma Concentration-time Curve From Time 0 to 2.5 Hours Postdose for Total Branched Chain Amino Acids (BCAA) Parameter in Cohorts 4a-2, 4b-2, 5a-2 and 5b-2
Time Frame: Day -1: pre-dose and Day 1 (2.5 hours post dose)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: micromole*hour per liter (mcmol*hr/L)
Arm/Group | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 2 | 5 | 2 | 6 | 2 | 6 | 2 | 6
micromole*hour per liter (mcmol*hr/L)
  Day-1: Total BCAA | 1257.10 (111.299) | 1372.16 (62.857) | 1125.05 (90.156) | 1102.43 (243.948) | 1879.40 (534.007) | 2124.73 (181.829) | 2011.75 (357.018) | 1982.10 (149.745)
  Day 1: Total BCAA | 1329.80 (64.912) | 1272.66 (84.565) | 1305.40 (172.393) | 1072.87 (178.282) | 2307.80 (568.514) | 1685.08 (163.129) | 2354.00 (433.174) | 1665.75 (119.524)

13. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Total BCAA Parameter in Cohorts 4a-2, 4b-2, 5a-2 and 5b-2
Time Frame: Day -1: pre-dose and Day 1 at multiple time points (0.5, 1, 1.5, 2, 2.5, 4, 5, 6, 10, 11, 12, 24 hours; up to 24 hours) post-dose
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 2 | 5 | 2 | 6 | 2 | 6 | 2 | 6
micromole per liter (mcmol/L)
  Day-1: Total BCAA | 603.85 (18.031) | 630.64 (21.031) | 483.00 (47.235) | 488.78 (112.097) | 938.00 (239.285) | 1161.05 (173.252) | 1027.25 (301.157) | 1072.32 (112.642)
  Day 1: Total BCAA | 604.90 (34.365) | 605.88 (60.406) | 593.25 (80.681) | 507.08 (85.660) | 1227.00 (386.222) | 800.78 (132.421) | 1227.65 (212.627) | 760.93 (48.105)

14. Secondary Outcome: Tmax: Time to Reach the Cmax for Total BCAA Parameter in Cohorts 4a-2, 4b-2, 5a-2 and 5b-2
Time Frame: as for outcome 13
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Number analyzed (Participants) | 2 | 5 | 2 | 6 | 2 | 6 | 2 | 6
hour
  Day-1: Total BCAA | 1.00 [1.0 to 1.0] | 1.00 [0.5 to 1.5] | 1.75 [1.0 to 2.5] | 0.75 [0.0 to 2.5] | 1.00 [1.0 to 1.0] | 1.00 [0.5 to 1.5] | 1.25 [1.0 to 1.5] | 1.00 [1.0 to 1.5]
  Day 1: Total BCAA | 1.00 [1.0 to 1.0] | 1.00 [0.5 to 1.0] | 1.75 [1.5 to 2.0] | 0.75 [0.5 to 1.0] | 1.00 [1.0 to 1.0] | 1.25 [1.0 to 2.0] | 1.00 [1.0 to 1.0] | 1.00 [0.5 to 2.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and up to Day 8.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1a-6a: Placebo | Cohort 1a: TAK-792 30 mg | Cohort 2a: TAK-792 100 mg | Cohort 3a: TAK-792 250 mg | Cohort 4a-1: TAK-792 500 mg | Cohort 5a-1: TAK-792 750 mg | Cohort 6a: TAK-792 1250 mg | Cohort 4a-2: Placebo | Cohort 4a-2: TAK-792 500 mg | Cohort 5a-2: Placebo | Cohort 5a-2: TAK-792 750 mg | Cohort 4b-1 - 6b: Placebo | Cohort 4b-1: TAK-792 500 mg | Cohort 5b-1: TAK-792 750 mg | Cohort 6b: TAK-792 1250 mg | Cohort 4b-2: Placebo | Cohort 4b-2: TAK-792 500 mg | Cohort 5b-2: Placebo | Cohort 5b-2: TAK-792 750 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/5 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 2/12 | 1/6 | 0/6 | 2/6 | 0/6 | 1/6 | 0/6 | 0/2 | 0/5 | 0/2 | 0/6 | 3/6 | 2/6 | 0/6 | 2/6 | 1/2 | 1/6 | 0/2 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a-6a: Placebo (N=12) | Cohort 1a: TAK-792 30 mg (N=6) | Cohort 2a: TAK-792 100 mg (N=6) | Cohort 3a: TAK-792 250 mg (N=6) | Cohort 4a-1: TAK-792 500 mg (N=6) | Cohort 5a-1: TAK-792 750 mg (N=6) | Cohort 6a: TAK-792 1250 mg (N=6) | Cohort 4a-2: Placebo (N=2) | Cohort 4a-2: TAK-792 500 mg (N=5) | Cohort 5a-2: Placebo (N=2) | Cohort 5a-2: TAK-792 750 mg (N=6) | Cohort 4b-1 - 6b: Placebo (N=6) | Cohort 4b-1: TAK-792 500 mg (N=6) | Cohort 5b-1: TAK-792 750 mg (N=6) | Cohort 6b: TAK-792 1250 mg (N=6) | Cohort 4b-2: Placebo (N=2) | Cohort 4b-2: TAK-792 500 mg (N=6) | Cohort 5b-2: Placebo (N=2) | Cohort 5b-2: TAK-792 750 mg (N=6)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.